CLINICAL TRIAL: NCT00844311
Title: Supplementation With hCG During Controlled Ovarian Stimulation With Recombinant FSH for in Vitro Fertilisation. A Randomized Controlled Clinical Study. Clinical, Embryological, Endocrine and Genetic Aspects.
Brief Title: Supplementation With Human Chorionic Gonadotropin (hCG) During Controlled Ovarian Stimulation With Recombinant Follicle-stimulating Hormone (FSH) for In Vitro Fertilisation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-257
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2009-02

CONDITIONS: Infertility
Keywords: hCG; human chorionic gonadotropin
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control arm (Active Comparator): 150 iu/day of rFSH alone
  Interventions: Drug: rFSH
- hCG low dose (Experimental): 150 iu/day of rFSH + 50 iu/day of hCG from stimulation day 1
  Interventions: Drug: rFSH; Drug: human chorionic gonadotropin
- hCG medium dose (Experimental): 150 iu/day of rFSH + 100 iu/day of hCG from stimulation day 1
  Interventions: Drug: rFSH; Drug: human chorionic gonadotropin
- hCG high dose (Experimental): 150 iu/day of rFSH + 150 iu/day of hCG from stimulation day 1
  Interventions: Drug: rFSH; Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: rFSH — 150 iu/day of rFSH
Drug: human chorionic gonadotropin — 50 iu/day of hCG from stimulation day 1
  Arms: hCG low dose
Drug: human chorionic gonadotropin — 100 iu/day of hCG from stimulation day 1
  Arms: hCG medium dose
Drug: human chorionic gonadotropin — 150 iu/day of hCG from stimulation day 1
  Arms: hCG high dose

SUMMARY:
The purpose of this trial is to study whether addition of different doses of human chorionic gonadotropins during controlled ovarian stimulation for patients undergoing IVF will improve the number of top-quality embryos.

ELIGIBILITY:
Inclusion Criteria:

1. Females with indication for COS and IVF;
2. Age between 25-37 years;
3. BMI >18 and < 30 kg/m2;
4. A regular menstrual cycle between 24 and 35 days and presumed to be ovulatory;
5. Two ovaries;
6. Tubal or unexplained infertility, including endometriosis stage I/II;
7. A uterus consistent with expected normal function (e.g. no clinically interfering uterine fibroids) documented by transvaginal ultrasound at the screening;
8. Male partner with sperm quality compatible with fertilization via IVF procedure or previous clinical pregnancy;
9. Early follicular phase serum FSH levels of 1-12 IU/l;
10. Early follicular phase total antral follicle (2-10mm) count ≥ 6;
11. Confirmation of down-regulation before randomisation by transvaginal ultrasound;
12. Willing and able to sign informed consent.

Exclusion Criteria:

1. History of or current PCOS, endometriosis stage III/IV or severe male factor requiring ICSI;
2. History of severe ovarian hyperstimulation syndrome (OHSS);
3. Presence of unilateral or bilateral hydrosalpinx at ultrasound;
4. More than three previously COS cycles;
5. Previous poor response on an IVF-cycle, defined as >20 days of gonadotrophin stimulation, cancellation due to limited follicular response or less than four follicles of ³15 mm diameter;
6. Previous IVF cycle with unsuccessful fertilization, defined as fertilisation of £20% of the retrieved oocytes;
7. History of recurrent miscarriage;
8. FSH>12IU/L or LH>12UI/L (early follicular phase);
9. Contraindications for the use of gonadotropins or GnRH analogues;
10. Recent history of current epilepsy, HIV infection, diabetes or cardiovascular gastrointestinal, hepatic, renal or pulmonary disease;
11. Pregnancy, lactation or contraindication to pregnancy;
12. Current past (last 12 months) abuse of alcohol or drugs;
13. History of chemotherapy (except for gestational conditions) of radiotherapy;
14. Undiagnosed vaginal bleeding;
15. Tumours of the ovary, breast, adrenal gland, pituitary or hypothalamus and malformation of sexual organs incompatible with pregnancy;
16. Abnormal karyotyping of the patient (if karyotyping is performed);
17. Hypersensitivity to any trial product.

Ages: 25 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Total number of top-quality embryos at day 3

SECONDARY OUTCOMES:
Implantation rate; Dose of rFSH needed; Serum levels of endocrine parameters; Ongoing pregnancy; Follicular fluid levels of endocrine parameters and cytokines; Expressions of gene families in granulosa cells and the cumulus complex.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Thuesen LL, Andersen AN, Loft A, Smitz J. Intrafollicular endocrine milieu after addition of hCG to recombinant FSH during controlled ovarian stimulation for in vitro fertilization. J Clin Endocrinol Metab. 2014 Feb;99(2):517-26. doi: 10.1210/jc.2013-1528. Epub 2013 Dec 2. PMID 24297796
- [Derived] Thuesen LL, Loft A, Egeberg AN, Smitz J, Petersen JH, Andersen AN. A randomized controlled dose-response pilot study of addition of hCG to recombinant FSH during controlled ovarian stimulation for in vitro fertilization. Hum Reprod. 2012 Oct;27(10):3074-84. doi: 10.1093/humrep/des256. Epub 2012 Jul 12. PMID 22791754